CLINICAL TRIAL: NCT00463593
Title: Schistosomiasis in Formal and Non-Formal Schools in Uganda: Implications for Control
Brief Title: Schistosomiasis in Formal and Non-Formal Schools in Uganda: Implications for Control Programmes
Status: Completed | Type: Observational
Sponsor: DBL -Institute for Health Research and Development (Other)
Other Study IDs: SRP-UG-NK-06
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Schistosomiasis; Helminthiasis; Anaemia
Keywords: schistosomiasis; helminthes; anaemia
MeSH Terms: conditions — Schistosomiasis; Helminthiasis; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — faeces blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: children enrolled in formal schools and children not enrolled in formal schools

SUMMARY:
Current efforts to control schistosomiasis and soil-transmitted helminthes infections focus on the school-age population, and school-based treatment delivery programs offer a major cost advantages because of the use of the existing school infrastructure and the fact that schoolchildren are accessible through schools. However, in many developing countries, large numbers of school-age children are not in school and this has raised questions about the effectiveness of school-based programs in reaching non-enrolled children. Increasingly, the non-formal education sector is providing a growing solution to the problem of poor enrolment in basic education, especially in sub-Saharan Africa, and has recently been used to deliver praziquantel as part of a national schistosomiasis control program in Uganda. However, it is unclear how effective this program has been in reaching children who attend non-formal schools and whether the program has been reaching children from the poorest households.

DETAILED DESCRIPTION:
This study will compare infection and nutritional status of children enrolled in formal schools and non-formal schools, and non-enrolled children in Nakasongola District in Uganda, and investigate the process and impact of treatment delivered by the national control program. The study will consist of household surveys and cross-sectional parasitological and hematological surveys, with follow-up six months later. The evaluation will take place over the course of a year and will:

* Compare the infection and nutritional status of children enrolled in formal schools and non-formal schools, and non-enrolled children in Nakasongola District, Uganda
* Compare programmatic process indicators, including enrolment rates, attendance rates, access to water and sanitation, treatment coverage in formal and non-formal schools
* Investigate the impact of treatment on intensity of infection and reinfection rates in formal and non-formal schools.

ELIGIBILITY:
Inclusion Criteria:

* School children in grad 1 and 2

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children enrolled in formal schools and children not enrolled in formal school identified by household survey
Sampling Method: Non-Probability Sample
Enrollment: 1293 (Actual)
Dates: Start 2006-12; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narcis Kabatereine, Dr, Principal Investigator — Vector Control Division, Ministry of Health Uganda
Locations (1):
- Vector Control Division, Kampala, Uganda